CLINICAL TRIAL: NCT05816421
Title: Reaching Optimal Implementation and Mental Health Outcomes for Underserved and Rural Communities in Foster and Kinship Care: Adaptation and Evaluation of the KEEP Model
Brief Title: Adaptation and Evaluation of the KEEP Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Stacey Tiberio, Principal Investigator, Oregon Social Learning Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R56MH129490 (NIH)
Record Dates: First submitted 2022-11-17; First posted 2023-04-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Depression, Anxiety; Post Traumatic Stress Disorder; Suicide and Self-harm; Externalizing Behavior
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Affinity KEEP (Experimental): Affinity KEEP groups are tailored to meet a specific population's needs and are comprised of parents who all share a common interest, purpose, or key characteristic. The four types of Affinity KEEP groups for this study include:
  * foster/kin parents of sexual and gender minority youth
  * foster/kin parents of Native youth
  * transracial placements where the youth and one or more parents are of a different race/ethnicity
  * groups delivered in Spanish
  Interventions: Behavioral: KEEP
- Non-Affinity KEEP (Active Comparator): Parents attending a Non-Affinity KEEP group.
  Interventions: Behavioral: Non-Affinity KEEP

INTERVENTIONS:
Behavioral: KEEP — The KEEP model focuses on optimizing the role of foster/kin parents as the agents of positive change for children and youth. Parent KEEP groups for children (ages 4-12) and KEEP-Safe groups for teens (ages 13-19) are delivered by two co-group leaders for 16 weeks. Sessions are 90 minutes each week. The same group of 8-10 foster/kin parents attends each week. Each KEEP group follows a manualized curriculum that emphasizes tailoring the content to the unique needs of the parents and youth in the group. The key parenting principles of the model include: (a) reinforce normative and prosocial behavior, (b) incentivize the behavior that parents want to promote, (c) build cooperation, (d) teach new behaviors, (e) use non-harsh effective limit setting, and (f) manage emotions while parenting.
  Arms: Affinity KEEP
Behavioral: Non-Affinity KEEP — Non-Affinity KEEP
  Arms: Non-Affinity KEEP

SUMMARY:
This study capitalizes on an opportunity to formally evaluate local adaptations of "Keeping Foster and Kinship Parents Supported and Trained" (KEEP), an evidence-based foster parent intervention, to reduce mental health disparities among child welfare-involved youth and improve care quality and long-term outcomes for Native, Hispanic/Latino, Black/African American, and sexual and gender minority youth. The knowledge gained from the study will impact all current and future large-scale implementations of KEEP and will bolster our scientific understanding the impact of KEEP on youth mental health outcomes.

DETAILED DESCRIPTION:
This study capitalizes on a contract with the Oregon Department of Human Services Child Welfare to implement KEEP state wide in Oregon with a focus on increasing access to services for minority youth populations. To help the child welfare system meet their goal of achieving health equity, adaptations to the KEEP curriculum have been made for minority groups, and KEEP is being delivered in "affinity groups". Affinity KEEP groups are tailored to meet a specific population's needs and are comprised of parents who all share a common interest, purpose, or key characteristic. To date, Affinity KEEP groups are being offered for foster/kin parents of populations defined by sexual and gender minority youth and Native youth, and for Spanish-speaking parents. The curriculum is currently being revised for transracial foster/kin placements where the youth and one or more parents are of a different race/ethnicity. The current proposal seeks to study N = 166 new families, as part of the ongoing Oregon KEEP implementation, and aggregate existing data from four KEEP studies to use propensity score matching to reduce selection bias and strengthen causal inferences that can be drawn from the potential benefits of providing KEEP to underserved minority populations. By leveraging two decades worth of data on the KEEP intervention and using state-of-the-art data harmonization techniques and a quasi-experimental design, this study affords a rigorous evaluation of whether tailoring the KEEP curriculum to minority populations' specific needs, and providing KEEP to foster/kin parents, improves youth mental health outcomes (i.e., depression/anxiety, post-traumatic stress disorder symptoms, suicidality, and externalizing behaviors) (Aim 1). The study could have a wide reach, impacting our understanding of how to improve and inform equitable delivery of services to youth and families involved in the child welfare system, and effectively address youth mental health disorders and improve care quality and long-term outcomes for a high-risk, underserved population of youth.

ELIGIBILITY:
Inclusion Criteria:

Foster/resource parents who have been recruited to attend KEEP and have a focal youth for the intervention that:

* is a dependent of Child Welfare Services in the state of Oregon
* is between the ages of 4 and 21 years.

Exclusion Criteria:

Foster/resource parents who have been recruited to attend KEEP and have a focal youth for the intervention that:

* is younger than 4 years of age.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 283 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Mean change in youth depression and anxiety symptoms | Baseline and 6-months post-baseline
  Psychometric scoring techniques will be used to harmonize items across multiple KEEP studies and instruments. Specifically, moderated nonlinear factor analysis will be utilized to estimate depression and anxiety symptoms factor scores that account for differential item functioning and impact across the set of study- and person-level covariates. Youth depression and anxiety symptoms will be measured via parent report using items from the Child Behavior Checklist and Parent Daily Report at baseline and 6-months post-baseline.
Mean change in youth post traumatic stress disorder (PTSD) symptoms | Baseline and 6-months post-baseline
  Psychometric scoring techniques will be used to harmonize items across multiple KEEP studies and instruments. Specifically, moderated nonlinear factor analysis will be utilized to estimate PTSD symptoms factor scores that account for differential item functioning and impact across the set of study- and person-level covariates. Youth PTSD symptoms will be measured via parent report using items from the Child Behavior Checklist and Parent Daily Report at baseline and 6-months post-baseline.
Mean change in youth self harming behaviors and suicidal ideation | Baseline and 6-months post-baseline
  Measured via parent report using the Child Behavior Checklist at baseline and 6-months post-baseline
Mean change in youth externalizing behaviors | Baseline and 6-months post-baseline
  Psychometric scoring techniques will be used to harmonize items across multiple KEEP studies and instruments. Specifically, moderated nonlinear factor analysis will be utilized to estimate externalizing behavior factor scores that account for differential item functioning and impact across the set of study- and person-level covariates. Youth externalizing behaviors will be measured via parent report using items from the Child Behavior Checklist and Parent Daily Report at baseline and 6-months post-baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Tiberio, PhD, Principal Investigator — Oregon Social Learning Center; Rohanna Buchanan, PhD, Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
These data will be archived with NIMH Data Archive.
URL: https://nda.nih.gov/edit_collection.html?id=4360